CLINICAL TRIAL: NCT01406626
Title: Effectiveness of Peer Navigation to Link Released HIV+ Jail Inmates to HIV Care
Acronym: LINK LA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Los Angeles County Department of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01DA030781 (NIH)
Record Dates: First submitted 2011-07-28; First posted 2011-08-01 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: HIV-infection/Aids
Keywords: HIV; AIDS; Peer navigation; Viral load; Corrections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peer Navigation Intervention Arm (Experimental): Subjects will receive the following peer navigation services:
  1) 10 Navigator meetings: Navigators will meet with participants in person to teach linkage/retention skills and knowledge
  2a) 2 Navigator accompaniment sessions: the peer navigator will accompany participants to HIV care appointment. Before and after the appointment, participants and navigators will review linkage and retention skills/knowledge and things that make it hard or easy for him/her to get regular HIV care
  2b) Optional peer navigator accompaniment sessions: If the participant requests, the peer navigator will provide accompaniment to supportive HIV care appointments (one per month max)
  3) 14 peer navigator care calls: During these calls, navigators and participants will talk about any problems that could make it difficult to get regular HIV care.
  Interventions: Behavioral: Peer Navigator
- Usual Care (No Intervention): Participants assigned to the control arm will receive the transitional case management (TCM) services that are currently offered at the jail

INTERVENTIONS:
Behavioral: Peer Navigator — Peer navigation intervention to improve linkage to and retention in HIV care and suppress viral load for underserved HIV+ persons in Los Angeles
  Arms: Peer Navigation Intervention Arm

SUMMARY:
This study will implement a peer navigation intervention to improve linkage to and retention in HIV care for inmates released from L.A. county jail into the community.

DETAILED DESCRIPTION:
The proposed study has two Primary Specific Aims:

1. To examine individual-level and structural-level barriers to HIV care after release from jail, using formative semi-structured interviews with ex-inmates, case managers, and HIV care providers; and to use the information we obtain to inform the adaptation and tailoring of an intervention designed to improve linkage with and retention to HIV care for HIV+ ex-inmates (Complete);
2. Using a two-group experimental RCT design, to test the adapted peer navigation intervention condition for HIV+ inmates upon release from jail compared to a usual care condition, and to evaluate the intervention's effectiveness at improving linkage with and retention in HIV care, self-reported ART adherence, and HIV RNA viral load suppression;

The intervention is hypothesized to result in greater linkage to care, a greater proportion completing at least three HIV care visits per year, increased self-reported ART adherence, and decreased levels of HIV RNA viral load compared to the usual care control group.

Secondary Aims of the study include assessing the potential moderating effects of substance abuse, the potential mediating effects of substance abuse treatment, and the program's effects on recidivism, and costs.

Active substance abuse is hypothesized to moderate the effect of the intervention, such that the intervention will be less effective among participants who report substance use.

ELIGIBILITY:
Inclusion criteria:

* Age 18 or older
* Men or TGW diagnosed HIV-positive
* English or bilingual Spanish speaking
* Selected for the TCM program (control condition) prior to LINK LA enrollment
* Residing in LA County upon release
* Eligible for ART or incarcerated on ART.

Exclusion criteria:

* Inability to give informed consent
* Parole hold or planned transfer to prison
* Stay in jail <5 days.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-represented transgender women.
Enrollment: 356 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Linkage to HIV Care | 12 months
  Number of HIV+ ex jail inmates accessing HIV care
Retention in Treatment | 12 months
  This assesses whether or not the HIV+ ex jail inmates were retained in their HIV care after first accessing care.
Adherence to Treatment | 12 months
  How adherent the HIV+ ex jail inmates are to their treatment regiment, by self-report.
Viral Load | 12 months
  HIV+ ex jail inmates' viral load

SECONDARY OUTCOMES:
Costs | 12 months
  Cost of the intervention and HIV care

CONTACTS AND LOCATIONS:
Overall Officials: William E Cunningham, MD, MPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- LA County Jail, Los Angeles, California, United States

REFERENCES:
- [Derived] Cunningham WE, Weiss RE, Nakazono T, Malek MA, Shoptaw SJ, Ettner SL, Harawa NT. Effectiveness of a Peer Navigation Intervention to Sustain Viral Suppression Among HIV-Positive Men and Transgender Women Released From Jail: The LINK LA Randomized Clinical Trial. JAMA Intern Med. 2018 Apr 1;178(4):542-553. doi: 10.1001/jamainternmed.2018.0150. PMID 29532059